CLINICAL TRIAL: NCT05764863
Title: fMRI Study of the Cerebal Bases of the Spatialization Process in Working Memory in Young Healthy Adults
Brief Title: fMRI Study of the Cerebal Bases of the Spatialization Process in Working Memory
Acronym: IRMF-SPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-PP-21
Record Dates: First submitted 2023-02-16; First posted 2023-03-13 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: One group of young healthy adults. Participants need to complete three experimental conditions associated with fMRI recording of brain activity. In condition A (Visual Spatial), participants will see the sequences presented from left to right; in condition B (Visual No Spatial), participants will see sequences of items presented in the middle of the screen; and in condition C (Auditory), the sequences will be presented in an auditory format.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- young healthy adults (Experimental): Participants need to complete three experimental conditions associated with fMRI recording of brain activity. In condition A (Visual Spatial), participants will see the sequences presented from left to right; in condition B (Visual No Spatial), participants will see sequences of items presented in the middle of the screen; and in condition C (Auditory), the sequences will be presented in an auditory format.
  Interventions: Radiation: fMRI

INTERVENTIONS:
Radiation: fMRI — The participant will then complete a series of working memory tasks under three distinct conditions as described above (visual spatial, visual non-spatial, auditory). The instructions and tasks will be administered via an MRI compatible monitor and headset system (NordicNeuroLab). During the tasks, the participant's brain activity will be recorded. Finally, at the end of the experiment, a high-resolution anatomical image of the brain will be acquired in order to facilitate the subsequent data processing steps and to define the position of the interparietal sulcus for each subject. The visit will be completed by a visual imaging questionnaire.

SUMMARY:
The present neuroimaging study investigates cerebral and behavioral markers of spatialization. Spatialization in memory corresponds to a mental representation of successive items from left to right in Westerners. A simple task to detect spatialization consists in presenting a series of stimuli sequentially. All stimuli are centered on the screen, so there is no spatial information during the task. After the presentation of the sequence, there is a recognition phase in which the participant is requested to take a decision as to whether a memory probe belongs to the sequence maintained in memory. The decision is made by pressing a key with the left or the right hand, depending on the instruction. The main measure is the difference in response times between the two hands. The standard spatialization effect in working memory in Westerners is that left-key responses are faster when retrieving the first items of the sequence whereas later items elicit faster right-key responses. To date, the factors that can influence this spatialization process in working memory as well as the brain structures involved remain largely unknown. Participants need to complete three experimental conditions associated with fMRI recording of brain activity. In task A (Visual Spatial), participants will see the sequences presented from left to right; in task B (Visual No Spatial), participants will see sequences of items presented in the middle of the screen; and in task C (Auditory), the sequences will be presented in an auditory format. When comparing tasks, A and B, we will be able to investigate if seeing information from left to right (spatialization is provided through the spatial coordinates of the items) is comparable to spatializing information from left to right (spatialization is not provided, all items have the same spatial coordinates). The comparison between task B and C will allow us to investigate the effect of seeing items (spatialization is not provided, all items have the same spatial coordinates) versus hearing them (spatialization is not provided and items have no spatial coordinates).

ELIGIBILITY:
Inclusion Criteria:

* right-handed adult subjects
* between 18 and 35 years of age,
* affiliated to or benefiting from a social security system
* having signed a prior informed consent.

Exclusion Criteria:

* minors
* subjects aged 36 years and older,
* left-handed,
* neurological disorders contraindicating fMRI examinations,
* protected by law under guardianship or curatorship, or unable to participate in a clinical study under Article L. 1121-16 of the French Public Health Code.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Behavioral measure | during the fMRI
  Reaction time (ms) across experimental conditions

SECONDARY OUTCOMES:
Brain measure | through study completion, an average of 2 years
  Brain activity recorded using fMRI device across experimental conditions
  level of Blood-Oxygen-Level-Dependant (BOLD) effect

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France